CLINICAL TRIAL: NCT00749580
Title: A Pilot, Randomized, Controlled Study to Evaluate the Safety and Efficacy of Raltegravir Versus NRTIs as a Backbone in HIV-Infected Patients Switched From a Stable Boosted PI Regimen
Brief Title: A Pilot,Raltegravir Versus NRTIs as a Backbone Switched From a Stable Boosted PI Regimen
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Florida (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); St. Joseph's Hospital, Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Merck-MK0518; NCT00717964 (obsolete NCT alias)
Record Dates: First submitted 2008-09-05; First posted 2008-09-09 (Estimated); Results first posted 2014-07-22 (Estimated); Last update posted 2014-12-17 (Estimated); Status verified 2014-06

CONDITIONS: Virus Diseases; HIV
Keywords: Safety
MeSH Terms: conditions — Virus Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1: Boosted PI+RAL (Experimental): Group 1 Raltegravir 400 mg PO b.i.d. + their current boosted PI regimen Subjects in this study are HIV-Infected Patients who are on a stable boosted PI regimen; in this group are assigned to switched from their NRTIs as a Backbone to Raltegravir
  Interventions: Drug: Switch NRTIs as a Backbone to Raltegravir
- 2: Boosted PI+NRTIs (No Intervention): Group 2 Continue the same regimen without change

INTERVENTIONS:
Drug: Switch NRTIs as a Backbone to Raltegravir — This is a multicenter, pilot randomized, controlled study to evaluate the safety and efficacy of raltegravir in patients switched from a stable boosted PI-based regimen with a NRTI backbone to raltegravir instead of their current NRTIs. A stable boosted PI-based regimen is defined as having a documented HIV RNA <75 copies/mL for ≥ 3 months prior to study entry, while receiving a boosted PI-based with NRTI backbone. Additionally, patients must not have had HIV RNA ≥ 75 copies/mL during the three months prior to study entry. Approximately 25 patients will be enrolled in the raltegravir treatment arm (Group 1) and approximately 25 patients in the continuation of the current NRTI backbone regimen treatment arm (Group 2). Patients will be randomly assigned 1:1 to a treatment group.
  Arms: 1: Boosted PI+RAL

SUMMARY:
The purpose of this study is to determine whether raltegravir 400 mg b.i.d. in a boosted PI regimen is as efficacious and safe as the NRTI backbone in a boosted PI regimen.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is a male or female at least 18 years of age on the day of signing the informed consent.
2. Patient is HIV positive as determined by enzyme-linked immunosorbent assay (ELISA) or HIV PCR.
3. Patient has documented HIV RNA <75 copies/mL for at least 3 months prior to study entry while on a stable boosted PI based regimen without a change in antiretroviral therapy and with no documentation of HIV RNA > or = 75 copies/mL during this time.
4. Patient has no history of documented coronary artery disease that clinical investigator deems as clinically significant.
5. Patient has the following laboratory values within 35 days prior to the treatment phase of this study:

   * Alkaline phosphatase ≤ 5.0 x upper limit of normal
   * AST (SGOT) and ALT (SGPT) ≤ 5.0 x upper limit of normal. Patients with Hepatitis C Coinfection may be enrolled provided the patients are stable and meet all eligibility criteria.
6. Patient has no clinical evidence of active pulmonary disease; at the investigators, discretion a chest x-ray could be obtained if felt necessary.
7. Patient who is of reproductive potential agrees to use an acceptable method of birth control throughout the study.
8. Patient agrees to remain off prohibited concomitant medications as outlined in Section 3.2.1 of the protocol.

Exclusion Criteria:

1. Patients who are currently failing a boosted PI based regimen.
2. Patient is receiving a second line boosted PI regimen including boosted tripranavir or boosted darunavir.
3. Patients with chronic hepatitis B infection.
4. Patient has a history or current evidence of any condition, therapy, laboratory abnormality or other circumstance that might confound the results of the study, or interfere with the patient's participation for the full duration of the study, such that it is not in the best interest of the patient to participate.
5. Patient has a history of alcohol or other substance abuse that in the opinion of the investigator would interfere with patient compliance or safety.
6. Patient is currently participating or has participated in a study with an investigational compound or device within 30 days of signing informed consent.
7. Patient has ever used any experimental HIV-integrase inhibitor.
8. Patient has used systemic immunosuppressive therapy (e.g., 20 mg or more of prednisone or equivalent per day) within one month prior to treatment in this study. Short courses of corticosteroids (e.g., as for asthma exacerbation) will be allowed.
9. Patient requires hemodialysis.
10. Patient has significant hypersensitivity or other contraindication to any of the components of the study drugs.
11. Patient has chronic hepatitis, including chronic hepatitis B and/or C and has decompensated liver disease.
12. Patient is pregnant or breastfeeding, or expecting to conceive (within the duration of the study). Patient is expecting to donate eggs (within the duration of the study). Patient is expecting to donate sperm (within the duration of the study).
13. Subjects who have received investigational medications within 30 days of baseline.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2008-11; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Hillsborough Health Department Specialty Care Center, Tampa, Florida, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the HIllsborough County Health Department, and Tampa Care Clinic, Tampa, Florida.
Pre-assignment Details: Per the inclusion and exclusion criteria
Groups:
- Switched: Group 1 Raltegravir 400 mg PO b.i.d. + their current boosted PI regimen
- Controlled: Group 2 Continue the same regimen without change
Period: Overall Study
Arm/Group | Switched | Controlled
Started | 21 (September 2008) | 25
Completed | 17 (December 2010) | 16
Not Completed | 4 | 9
Not completed — Lost to Follow-up | 4 | 8
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- 1: Boosted PI+RAL: Group 1 Raltegravir 400 mg PO b.i.d. + their current boosted PI regimen
- Total: Total of all reporting groups
Arm/Group | 1: Boosted PI+RAL | 2: Boosted PI+NRTIs | Total
Number analyzed (Participants) | 21 | 25 | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 25 | 46
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (9) | 49 (8) | 47 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 15 | 19 | 34
Region of Enrollment [Number; unit: participants]
  United States | 21 | 25 | 46

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Suppressed Viral Load(<75 Copies/ml)in Raltegravir 400 mg Bid vs. NRTI Backbone, Each in Combination of Boosted PI Regimen
Description: Number of patients with virologic suppression< 75 copies/ ml at 24 wk,in raltegravir 400 mg bid vs. NRTI backbone, each in combination of boosted PI regimen.
Time Frame: at 24weeks for each patient
Measure: Number; unit: participants
Groups:
- Boosted PI+RAL: Switch NRTI backbone to RAL
- Boosted PI+NRTIs: Continue the same regimen without change
Arm/Group | Boosted PI+RAL | Boosted PI+NRTIs
Number analyzed (Participants) | 21 | 19
participants | 18 | 18
Statistical Analysis 1: Comparison: Boosted PI+RAL vs Boosted PI+NRTIs; Test type: Superiority or Other; p = 0.935, Fisher Exact

2. Secondary Outcome: Virologic Suppression of < 75 Copies/ml at 48 Weeks
Time Frame: at 48 weeks for each patient
Measure: Number; unit: participants
Arm/Group | Boosted PI+RAL | Boosted PI+NRTIs
Number analyzed (Participants) | 17 | 17
participants | 14 | 16

ADVERSE EVENTS:
Arm/Group | Switched | Controlled
Serious Adverse Events (participants affected / at risk) | 0/21 | 1/25
Other Adverse Events (participants affected / at risk) | 18/21 | 18/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Switched (N=21) | Controlled (N=25)
Faconi syndrome (Renal and urinary disorders) | 0 | 1 — Faconi's syndrome in a patient who is on TDF/FTC base regimen. The patient recovered, the regimen switched TDF/FTC was switched to TDF sparing regimen and the patient was wihtdrawn form the study.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Switched (N=21) | Controlled (N=25)
Erthema (Skin and subcutaneous tissue disorders) | 1 | 1 — Grade 1, Not related, not anticipated
Constipation (Gastrointestinal disorders) | 2 | 3 — Grade 1, Not related, not anticipated
Pruritus( local, not drug rash)) (Skin and subcutaneous tissue disorders) | 2 | 1 — Grade 1, Not related, not anticipated
fatigue (General disorders) | 1 | 2 — Grade 1, Not related, not anticipated
swelling (Skin and subcutaneous tissue disorders) | 2 | 0 — Grade 2, Not related, not anticipated
rash (Skin and subcutaneous tissue disorders) | 1 | 1 — Grade 1, Not related, not anticipated
Instability (Nervous system disorders) | 1 | 0 — Grade 2, Not related, not anticipated
loss appetitie (General disorders) | 0 | 2 — Grade 1, Not related, not anticipated
Headache (Nervous system disorders) | 6 | 1 — Grade 1, Not related, and anticipated Two event in the RAL arm is grade 2. Not related, and anticipated
Depression (Psychiatric disorders) | 1 | 0 — Grade 1, Not related, not anticipated
Insomnia (Psychiatric disorders) | 0 | 1 — Grade 1, Not related, not anticipated
dry mouth (General disorders) | 2 | 0 — Grade 1, Not related, not anticipated
wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 — Grade 1, Not related, not anticipated
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 — Grade 1, Not related, not anticipated
Worsening seasonal allergy (Immune system disorders) | 0 | 1 — Grade 1, Not related, not anticipated
sore throat (Infections and infestations) | 1 | 0 — Grade 1, Not related, not anticipated
weight gain (General disorders) | 1 | 0 — Grade 1, Not related, not anticipated
vomiting (Gastrointestinal disorders) | 1 | 1 — Grade 2, Not related, not anticipated
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 — Grade 1, Not related, not anticipated
Urinary frequency (Renal and urinary disorders) | 1 | 0 — Grade 1, Not related, not anticipated
flatulence (Gastrointestinal disorders) | 1 | 0 — Grade 1, Not related, not anticipated
Increase appetite (General disorders) | 1 | 0 — Grade 1, Not related, not anticipated
Dizziness (General disorders) | 1 | 0 — Grade 1, Not related, not anticipated
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 | 1 — Grade 1 and 2, Not related, not anticipated
abdominal pain (Gastrointestinal disorders) | 0 | 1 — Grade 2, Not related, not anticipated
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 — Grade 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 — Grade 2
Condyloma removal (Surgical and medical procedures) | 1 | 0 — Grade 2-not related
Squamous cell carcinoma insitu (Skin and subcutaneous tissue disorders) | 1 | 0 — Grade 2-not related
diarrhea (Gastrointestinal disorders) | 0 | 1 — Grade 1
Abnormal liver function (Gastrointestinal disorders) | 1 | 0 — Grade 3, recovered , no action taken
Basal cell carcinoma (Skin and subcutaneous tissue disorders) | 1 | 0 — Grade 1-no action taken

LIMITATIONS AND CAVEATS:
This is a pilot study and has a small sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No